CLINICAL TRIAL: NCT04010227
Title: Telephone Support for Advanced Gastrointestinal Cancer Patients and Their Family Caregivers
Brief Title: Telephone Support for Advanced Gastrointestinal Cancer Patients and Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Catherine Mosher, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1904388865; R21CA235788 (NIH)
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Results first posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-11

CONDITIONS: Gastrointestinal Neoplasms
Keywords: Acceptance and Commitment Therapy; Fatigue; Family Caregivers; Psychotherapy
MeSH Terms: conditions — Gastrointestinal Neoplasms; Fatigue | interventions — Acceptance and Commitment Therapy; Educational Status; Palliative Care

STUDY DESIGN:
Intervention Model Description: Advanced gastrointestinal cancer patient-family caregiver dyads (N = 40) were randomly assigned in equal numbers to Acceptance and Commitment Therapy (ACT) or education/support using a stratified block randomization scheme to balance the groups by patient performance status (patient-reported Eastern Cooperative Oncology Group [ECOG] scores 0 or 1 vs. 2).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and Commitment Therapy (Experimental): Patients and caregivers in the ACT arm learn new and more adaptive ways to respond to difficult internal experiences (e.g., fatigue, thoughts, and feelings).
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Education/Support (Active Comparator): Patients and caregivers in the education/support arm discuss their cancer-related concerns and receive education on services available in their medical center and community.
  Interventions: Behavioral: Education/Support

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Across six weekly 50-minute sessions, advanced GI cancer patients and caregivers practice various mindfulness exercises, clarify their values, and set specific goals in alignment with their values. Through in-session and home practice of skills, participants learn new and more adaptive ways to respond to unwanted internal experiences (e.g., fatigue, distress). Participants receive handouts on session topics and a compact disc (CD) that we developed to guide mindfulness practices.
  Arms: Acceptance and Commitment Therapy
Behavioral: Education/Support — Across six weekly 50-minute sessions, advanced GI cancer patients and caregivers are directed to resources for practical and health information and contact information for psychosocial services. Sessions include an orientation to the patient's medical center and treatment team, education regarding common quality-of-life concerns experienced by cancer patients and caregivers, and an overview of medical center and community resources for addressing these concerns. The therapist also describes resources for addressing financial concerns and methods of evaluating health information available via the Internet and other modalities. Participants receive handouts summarizing session topics and are asked to review them as homework.
  Arms: Education/Support

SUMMARY:
This trial tests telephone-based Acceptance and Commitment Therapy (ACT), a type of psychotherapy, to reduce fatigue interference with activities, mood, and cognition in advanced gastrointestinal (GI) cancer patients and family caregiver burden. ACT includes mindfulness exercises (e.g., meditations, performing activities with greater awareness), identifying personal values (e.g., family, spirituality), and engaging in activities consistent with these values. A total of 40 patient-caregiver dyads were randomly assigned in equal numbers to either the ACT intervention or an education/support condition. Dyads in both conditions participated in six weekly 50-minute telephone sessions. Outcomes were assessed at baseline, 2 weeks post-intervention, and 3 months post-intervention. The investigators hypothesize that ACT will lead to improved primary and secondary outcomes as compared to education/support. Study findings will inform a large-scale trial of intervention efficacy.

DETAILED DESCRIPTION:
This trial evaluates the feasibility, acceptability, and preliminary efficacy of telephone-based Acceptance and Commitment Therapy (ACT) on fatigue interference in advanced gastrointestinal (GI) cancer patients and family caregiver burden as well as secondary outcomes. The study team recruited advanced GI cancer patients receiving care at the Indiana University Simon Cancer Center or Eskenazi Health hospital. Potentially eligible patients were mailed an introductory letter signed by their oncologist and the PI along with a consent form. The letter had a number to call if they did not wish to be contacted further. A research assistant (RA) called all prospective participants who did not opt out approximately 1 to 2 weeks after the letter was mailed. The RA described the study as outlined in the consent form and answered any questions. Then the RA administered an eligibility screening to those who consented to participate. Eligible and consenting patients identified a potentially eligible family caregiver. If the family caregiver was eligible and consented to participate, then the patient and caregiver each completed a baseline phone assessment. Following baseline assessments, patient-caregiver dyads (N = 40 dyads) were randomly assigned in equal numbers to ACT or education/support using a stratified block randomization scheme to balance the groups by patient performance status (patient-reported Eastern Cooperative Oncology Group [ECOG] scores 0 or 1 vs. 2). Dyads in both study conditions completed six weekly 50-minute telephone sessions with the first session occurring one week after baseline. For ACT participants, adherence to home practice during the past week was assessed and recorded during each session. Feasibility will be examined via accrual, attrition, and adherence rates, and acceptability will be evaluated using a mixed methods approach (qualitative and quantitative). Blind interviewers assessed outcomes during follow-up phone assessments at 2 weeks and 3 months post-intervention.

ELIGIBILITY:
Patient Inclusion Criteria:

* Patient is at least 3 weeks post-diagnosis of unresectable stage III or stage IV gastrointestinal cancer (i.e., anal, colon, esophageal, gallbladder, liver, pancreatic, rectal, small intestine, or stomach cancer) and is receiving care at the Indiana University Simon Cancer Center or Eskenazi Health.
* Patient is at least 21 years of age.
* Patient can speak and read English.
* Patient has an eligible, consenting family caregiver (see criteria below).
* Patient has moderate to severe fatigue interference with functioning.

Patient Exclusion Criteria:

* Patient shows significant psychiatric or cognitive impairment that would preclude providing informed consent and study participation.
* Patient reports being able to do little activity on a functional status measure.
* Patient is receiving hospice care at screening.
* Patient does not have working phone service.
* Patient has hearing impairment that precludes participation.

Caregiver Inclusion Criteria:

* Family caregiver identified by a stage IV gastrointestinal cancer patient who meets the eligibility criteria.
* Caregiver has significant caregiving burden or distress
* Caregiver lives with the patient or has visited the patient in-person at least twice a week for the past month.
* Caregiver is at least 18 years of age.
* Caregiver can speak and read English.

Caregiver Exclusion Criteria:

* Caregiver shows significant psychiatric or cognitive impairment that would preclude providing informed consent and study participation.
* Caregiver does not have working phone service.
* Caregiver has hearing impairment that precludes participation.
* Patient declines study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine E Mosher, Ph.D., Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Eskenazi Health, Indianapolis, Indiana
  - Indiana University Simon Comprehensive Cancer Center, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: Yes
Results of this trial will be presented at professional meetings and published in peer-reviewed journals. The data set will be made available to qualified investigators within 6 months of the publication of the primary outcome paper. The data set will contain necessary identifiers, excluding those prohibited by HIPAA. The investigators will be required to sign a data use agreement and obtain Institutional Review Board (IRB) approval before receiving the data set.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data set will be made available to qualified investigators within 6 months of the publication of the primary outcome paper. Data will be available for at least 6 years.
Access Criteria: The data set and supporting information will be made available to qualified investigators to allow replication of analyses or secondary data analyses. The PI will review requests for data access. The investigators will be required to sign a data use agreement and obtain IRB approval before receiving the data set. The mechanism for data sharing will be reviewed by the IRB.

REFERENCES:
- [Background] Mosher CE, Secinti E, Kroenke K, Helft PR, Turk AA, Loehrer PJ Sr, Sehdev A, Al-Hader AA, Champion VL, Johns SA. Acceptance and commitment therapy for fatigue interference in advanced gastrointestinal cancer and caregiver burden: protocol of a pilot randomized controlled trial. Pilot Feasibility Stud. 2021 Apr 20;7(1):99. doi: 10.1186/s40814-021-00837-9. PMID 33879253
- [Result] Mosher CE, Secinti E, Wu W, Kashy DA, Kroenke K, Bricker JB, Helft PR, Turk AA, Loehrer PJ, Sehdev A, Al-Hader AA, Champion VL, Johns SA. Acceptance and commitment therapy for patient fatigue interference and caregiver burden in advanced gastrointestinal cancer: Results of a pilot randomized trial. Palliat Med. 2022 Jul;36(7):1104-1117. doi: 10.1177/02692163221099610. Epub 2022 May 30. PMID 35637615

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 patients and 2 caregivers were excluded from the study before assignment to groups. Here is a list of the reasons:
  Patient death (1) Caregiver withdrew because patient died (1) Patient lost to follow-up (1) Caregiver withdrew because patient was lost to follow-up (1)
Groups:
- Acceptance and Commitment Therapy: Patients and caregivers in the Acceptance and Commitment Therapy arm learn new and more adaptive ways to respond to difficult internal experiences (e.g., fatigue, thoughts, and feelings).
  Acceptance and Commitment Therapy: Across six weekly 50-minute sessions, advanced GI cancer patients and caregivers practice various mindfulness exercises, clarify their values, and set specific goals in alignment with their values. Through in-session and home practice of skills, participants learn new and more adaptive ways to respond to unwanted internal experiences (e.g., fatigue, distress). Participants receive handouts on session topics and a compact disc (CD) that we developed to guide mindfulness practices.
Period: Overall Study
Arm/Group | Acceptance and Commitment Therapy | Education/Support
Started | 40 | 40
Patients Started | 20 | 20
Caregivers Started | 20 | 20
Completed | 28 | 30
Not Completed | 12 | 10
Not completed — Death | 1 | 2
Not completed — Medical Reasons | 4 | 3
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Caregiver withdrawn because patient was withdrawn for any reason | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Acceptance and Commitment Therapy: Patients and caregivers in the ACT arm learn new and more adaptive ways to respond to difficult internal experiences (e.g., fatigue, thoughts, and feelings).
  Acceptance and Commitment Therapy: Across six weekly 50-minute sessions, advanced GI cancer patients and caregivers practice various mindfulness exercises, clarify their values, and set specific goals in alignment with their values. Through in-session and home practice of skills, participants learn new and more adaptive ways to respond to unwanted internal experiences (e.g., fatigue, distress). Participants receive handouts on session topics and a CD that we developed to guide mindfulness practices.
- Total: Total of all reporting groups
Arm/Group | Acceptance and Commitment Therapy | Education/Support | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] — Patient and caregiver age Population: Age data are presented separately for patients and caregivers.
  years
    Patient age: number analyzed (Participants) | 20 | 20 | 40
    Patient age | 59.25 (9.96) | 57.85 (15.71) | 58.55 (13.00)
    Caregiver age: number analyzed (Participants) | 20 | 20 | 40
    Caregiver age | 55.55 (14.87) | 48.60 (15.80) | 52.08 (15.55)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex data are presented separately for patients and caregivers.
  Participants
    Patient age: number analyzed (Participants) | 20 | 20 | 40
    Patient age: Female | 10 | 8 | 18
    Patient age: Male | 10 | 12 | 22
    Caregiver age: number analyzed (Participants) | 20 | 20 | 40
    Caregiver age: Female | 3 | 7 | 10
    Caregiver age: Male | 17 | 13 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 40 | 40 | 80
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Racial data are presented separately for patients and caregivers.
  Participants
    Patient race: number analyzed (Participants) | 20 | 20 | 40
    Patient race: American Indian or Alaska Native | 0 | 0 | 0
    Patient race: Asian | 0 | 0 | 0
    Patient race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Patient race: Black or African American | 1 | 1 | 2
    Patient race: White | 19 | 19 | 38
    Patient race: More than one race | 0 | 0 | 0
    Patient race: Unknown or Not Reported | 0 | 0 | 0
    Caregiver race: number analyzed (Participants) | 20 | 20 | 40
    Caregiver race: American Indian or Alaska Native | 0 | 0 | 0
    Caregiver race: Asian | 0 | 0 | 0
    Caregiver race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Caregiver race: Black or African American | 2 | 1 | 3
    Caregiver race: White | 18 | 19 | 37
    Caregiver race: More than one race | 0 | 0 | 0
    Caregiver race: Unknown or Not Reported | 0 | 0 | 0
Fatigue Interference Subscale of Fatigue Symptom Inventory [Mean (Standard Deviation); unit: units on a scale] — Seven items are rated on 11-point scales (0=no interference to 10=extreme interference) that assess the extent to which fatigue in the past week interfered with general level of activity, ability to bathe and dress, normal work activity (including housework), ability to concentrate, relations with others, enjoyment of life, and mood. The seven items are summed with higher total scores indicating greater fatigue interference. The total score range is 0 to 70. This is the primary outcome for patients. Population: This outcome was only collected on patients.
  units on a scale
    number analyzed (Participants) | 20 | 20 | 40
    (all) | 4.25 (1.86) | 3.58 (1.92) | 3.91 (1.90)
Short-Form of Zarit Burden Interview [Mean (Standard Deviation); unit: units on a scale] — Twelve items are rated on 5-point scales (0=never to 4=nearly always) that assess personal strain and role strain due to caregiving. The 12 items are summed with higher total scores indicating greater caregiving burden. The total score range is 0 to 48. This is the primary outcome for caregivers. Population: This primary outcome measure was only collected on caregivers.
  units on a scale
    number analyzed (Participants) | 20 | 20 | 40
    (all) | 15.85 (3.82) | 18.45 (8.52) | 17.15 (6.65)
Education [Mean (Standard Deviation); unit: years] — Years of education Population: Education data are presented separately for patients and caregivers.
  years
    Patient education: number analyzed (Participants) | 20 | 20 | 40
    Patient education | 15.48 (2.66) | 14.70 (2.45) | 15.09 (2.56)
    Caregiver education: number analyzed (Participants) | 20 | 20 | 40
    Caregiver education | 15.23 (2.67) | 15.45 (2.61) | 15.34 (2.61)
Household income [Count of Participants; unit: Participants] — Income data were collected in categories. Population: Income data are presented separately for patients and caregivers.
  Participants
    Patient income: number analyzed (Participants) | 20 | 20 | 40
    Patient income: $0-$50,999 | 5 | 7 | 12
    Patient income: $51,000-$99,999 | 5 | 3 | 8
    Patient income: $100,000 or more | 10 | 9 | 19
    Patient income: Missing data | 0 | 1 | 1
    Caregiver income: number analyzed (Participants) | 20 | 20 | 40
    Caregiver income: $0-$50,999 | 5 | 6 | 11
    Caregiver income: $51,000-$99,999 | 9 | 5 | 14
    Caregiver income: $100,000 or more | 6 | 9 | 15
    Caregiver income: Missing data | 0 | 0 | 0
Caregiver's relationship to the patient [Count of Participants; unit: Participants] — Population: Data are specific to caregivers.
  Participants
    number analyzed (Participants) | 20 | 20 | 40
    Spouse or partner | 12 | 13 | 25
    Other family member | 8 | 7 | 15
Caregiver lives with the patient [Count of Participants; unit: Participants] — Population: Data are specific to caregivers.
  Participants
    number analyzed (Participants) | 20 | 20 | 40
    Yes, caregiver lives with the patient. | 15 | 15 | 30
    No, caregiver does not live with the patient. | 5 | 5 | 10
Type of gastrointestinal cancer [Count of Participants; unit: Participants] — Collected from patient medical records Population: Data are specific to patients.
  Participants
    number analyzed (Participants) | 20 | 20 | 40
    Colorectal cancer | 10 | 6 | 16
    Pancreatic cancer | 3 | 7 | 10
    Other gastrointestinal cancer | 7 | 7 | 14
Time since gastrointestinal cancer diagnosis [Mean (Standard Deviation); unit: years] — Collected from patient medical records at baseline Population: Data are specific to patients.
  years
    number analyzed (Participants) | 20 | 20 | 40
    (all) | 2.40 (2.36) | 1.67 (3.30) | 2.04 (2.85)
Chemotherapy [Count of Participants; unit: Participants] — Collected from patient medical records at baseline Population: Data are specific to patients.
  Participants
    number analyzed (Participants) | 20 | 20 | 40
    Yes-chemotherapy received for gastrointestinal cancer | 15 | 17 | 32
    No-chemotherapy not received for gastrointestinal cancer | 5 | 3 | 8
Radiation [Count of Participants; unit: Participants] — Data collected from patient medical records at baseline. Population: Data are specific to patients.
  Participants
    number analyzed (Participants) | 20 | 20 | 40
    Yes-radiation received for gastrointestinal cancer | 2 | 6 | 8
    No-radiation not received for gastrointestinal cancer | 18 | 14 | 32
Chemoradiation [Count of Participants; unit: Participants] — Data collected from patient medical records at baseline. Population: Data are specific to patients.
  Participants
    number analyzed (Participants) | 20 | 20 | 40
    Yes-chemoradiation received for gastrointestinal cancer | 5 | 4 | 9
    No-chemoradiation not received for gastrointestinal cancer | 15 | 16 | 31
Surgery to remove primary tumor [Count of Participants; unit: Participants] — Data were collected from patient medical records at baseline. Population: Data are specific to patients.
  Participants
    number analyzed (Participants) | 20 | 20 | 40
    Yes-surgery received to remove primary tumor | 12 | 11 | 23
    No-surgery not received to remove primary tumor | 8 | 9 | 17
Surgery to remove metastases [Count of Participants; unit: Participants] — Data were collected from patient medical records at baseline. Population: Data are specific to patients.
  Participants
    number analyzed (Participants) | 20 | 20 | 40
    Yes-received surgery to remove metastases | 7 | 4 | 11
    No--did not receive surgery to remove metastases | 13 | 16 | 29
Targeted Therapy [Count of Participants; unit: Participants] — Data were collected from patient medical records at baseline. Population: Data are specific to patients.
  Participants
    number analyzed (Participants) | 20 | 20 | 40
    Yes, received targeted therapy for gastrointestinal cancer | 9 | 5 | 14
    No, did not receive targeted therapy for gastrointestinal cancer | 11 | 15 | 26

OUTCOME MEASURES:

1. Primary Outcome: Fatigue Interference Subscale of Fatigue Symptom Inventory
Description: Seven items are rated on 11-point scales (0=no interference to 10=extreme interference) that assess the extent to which fatigue in the past week interfered with general level of activity, ability to bathe and dress, normal work activity (including housework), ability to concentrate, relations with others, enjoyment of life, and mood. The seven items are summed with higher total scores indicating greater fatigue interference. The total score range is 0 to 70. This is the primary outcome for patients.
Time Frame: 2 weeks and 3 months post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acceptance and Commitment Therapy | Education/Support
Number analyzed (Participants) | 20 | 20
units on a scale
  Patient fatigue interference at 2 weeks post-intervention | 3.93 (2.17) | 3.47 (2.54)
  Patient fatigue interference at 3 months post-intervention | 4.27 (1.66) | 4.26 (2.12)
Statistical Analysis 1: Comparison: Acceptance and Commitment Therapy vs Education/Support; Test type: Superiority; p = 0.60, Mixed Models Analysis — P-value for study group x time interaction. Two-tailed p-values <.05 were considered statistically significant; degrees of freedom = 76. multiply imputed data were used in analyses; partial correlation = 0.08, 95% CI 2-sided [-0.23 to 0.40]

2. Primary Outcome: Short-form of Zarit Burden Interview
Description: Twelve items are rated on 5-point scales (0=never to 4=nearly always) that assess personal strain and role strain due to caregiving. The 12 items are summed with higher total scores indicating greater caregiving burden. The total score range is 0 to 48. This is the primary outcome for caregivers.
Time Frame: 2 weeks and 3 months post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acceptance and Commitment Therapy | Education/Support
Number analyzed (Participants) | 20 | 20
units on a scale
  Caregiver burden at 2 weeks post-intervention | 13.92 (3.86) | 16.37 (7.10)
  Caregiver burden at 3 months post-intervention | 15.32 (4.59) | 18.17 (8.36)
Statistical Analysis 1: Comparison: Acceptance and Commitment Therapy vs Education/Support; Test type: Superiority; p = 0.96, Mixed Models Analysis — P-value for study group x time interaction. Two-tailed p-values <.05 were considered statistically significant; degrees of freedom = 76. Multiply imputed data were used; partial correlation = 0.02, 95% CI 2-sided [-0.29 to 0.34]

3. Secondary Outcome: Patient-Reported Outcome Measurement Information System (PROMIS) Sleep-Related Impairment
Description: This 8-item measure assesses the perceived interference of sleep problems with activities, mood, and cognition (e.g., difficulty concentrating or completing tasks). Each item is rated on a scale from 1 (not at all) to 5 (very much). Item #2 is reverse-scored and then the 8 items are summed with higher total scores indicating greater sleep-related impairment. The total scores are converted to T-scores with a range from 30.0 to 80.1. Higher T-scores indicate a worse outcome. The population mean for T-scores is 50 with a standard deviation of 10. This is a secondary outcome for patients.
Time Frame: 2 weeks and 3 months post-intervention
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Acceptance and Commitment Therapy | Education/Support
Number analyzed (Participants) | 20 | 20
T-score
  Patient sleep-related impairment at 2 weeks post-intervention | 57.37 (4.03) | 52.99 (8.38)
  Patient sleep-related impairment at 3 months post-intervention | 56.91 (5.22) | 53.86 (7.41)
Statistical Analysis 1: Comparison: Acceptance and Commitment Therapy vs Education/Support; Test type: Superiority; p = 0.75, Mixed Models Analysis — P-value for study group x time interaction. Two-tailed p-values <.05 were considered statistically significant; degrees of freedom = 76. Multiply imputed data were used; partial correlation = 0.06, 95% CI 2-sided [-0.25 to 0.38]

4. Secondary Outcome: PROMIS Ability to Participate in Social Roles and Activities
Description: This 6-item measure assesses participants' ability to participate in social roles and activities. The items measure difficulty engaging in social and recreational activities as well as usual work (including housework). Each item is rated on a scale from 1 (never) to 5 (always) and is reverse coded. Then the six items are summed with higher total scores indicating greater ability to participate in social roles and activities. The total scores are converted to T-scores with a range from 26.7 to 65.0 with higher scores indicating a better outcome. The population mean for T-scores is 50 with a standard deviation of 10. This is a secondary outcome for both patients and caregivers.
Time Frame: 2 weeks and 3 months post-intervention
Population: Number analyzed = 20 patients and 20 caregivers in the Acceptance and Commitment Therapy arm and 20 patients and 20 caregivers in the Education/Support arm
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Acceptance and Commitment Therapy | Education/Support
Number analyzed (Participants) | 40 | 40
T-score
  Patient ability to participate in social roles and activities at 2 weeks post-intervention: number analyzed (Participants) | 20 | 20
  Patient ability to participate in social roles and activities at 2 weeks post-intervention | 45.02 (6.60) | 42.42 (7.26)
  Patient ability to participate in social roles and activities at 3 months post-intervention: number analyzed (Participants) | 20 | 20
  Patient ability to participate in social roles and activities at 3 months post-intervention | 45.58 (6.92) | 46.14 (5.01)
  Caregiver ability to participate in social roles and activities at 2 weeks post-intervention: number analyzed (Participants) | 20 | 20
  Caregiver ability to participate in social roles and activities at 2 weeks post-intervention | 42.56 (4.66) | 40.40 (7.05)
  Caregiver ability to participate in social roles and activities at 3 months post-intervention: number analyzed (Participants) | 20 | 20
  Caregiver ability to participate in social roles and activities at 3 months post-intervention | 40.34 (2.62) | 41.04 (8.11)
Statistical Analysis 1: Comparison: Acceptance and Commitment Therapy vs Education/Support; Test type: Superiority; p = 0.33, Mixed Models Analysis — P-value for study group x time interaction. Two-tailed p-values <.05 were considered statistically significant; degrees of freedom = 144. Multiply imputed data were used; partial correlation = 0.09, 95% CI 2-sided [-0.23 to 0.40]

5. Secondary Outcome: Acceptance and Action Questionnaire-II
Description: This 7-item measure assesses psychological flexibility, or the ability to fully experience the present moment while persisting in actions aligned with personal values. Each item is rated on a scale from 1 (never true) to 7 (always true). The seven items are summed with higher total scores indicating greater levels of psychological inflexibility. The total score range is 7 to 49. This is a secondary outcome for both patients and caregivers.
Time Frame: 2 weeks and 3 months post-intervention
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acceptance and Commitment Therapy | Education/Support
Number analyzed (Participants) | 40 | 40
units on a scale
  Patient psychological inflexibility at 2 weeks post-intervention: number analyzed (Participants) | 20 | 20
  Patient psychological inflexibility at 2 weeks post-intervention | 13.82 (4.98) | 14.52 (6.45)
  Patient psychological inflexibility at 3 months post-intervention: number analyzed (Participants) | 20 | 20
  Patient psychological inflexibility at 3 months post-intervention | 13.85 (6.04) | 15.97 (5.61)
  Caregiver psychological inflexibility at 2 weeks post-intervention: number analyzed (Participants) | 20 | 20
  Caregiver psychological inflexibility at 2 weeks post-intervention | 17.77 (6.45) | 17.45 (8.22)
  Caregiver psychological inflexibility at 3 months post-intervention: number analyzed (Participants) | 20 | 20
  Caregiver psychological inflexibility at 3 months post-intervention | 17.58 (6.21) | 17.79 (6.41)
Statistical Analysis 1: Comparison: Acceptance and Commitment Therapy vs Education/Support; Test type: Superiority; p = 0.91, Mixed Models Analysis — P-value for study group x time interaction. Two-tailed p-values <.05 were considered statistically significant; degrees of freedom = 144. Multiply imputed data were used; partial correlation = 0.03, 95% CI 2-sided [-0.29 to 0.34]

6. Secondary Outcome: McGill Quality of Life Questionnaire-Revised
Description: This 15-item measure evaluates physical, psychological, existential, and social quality of life in patients with serious illnesses. Each of the 4 subscale scores (i.e., physical, psychological, existential, and social quality of life) is the sum of the items with higher scores indicating better quality of life. Items are rated on 0 to 10 scales. The physical quality of life subscale is the sum of 3 items (2 items reverse-coded) with a range of 0 to 30. The psychological quality of life subscale is the sum of 4 items (all items reverse-coded) with a range of 0 to 40. The existential quality of life subscale is the sum of 4 items (1 item reverse-coded) with a range of 0 to 40. The social quality of life subscale is the sum of 3 items (none reverse-coded) with a range of 0 to 30. This is a secondary outcome measure for patients.
Time Frame: 2 weeks and 3 months post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acceptance and Commitment Therapy | Education/Support
Number analyzed (Participants) | 20 | 20
units on a scale
  Patient physical quality of life at 2 weeks post-intervention | 17.30 (6.34) | 16.89 (6.20)
  Patient physical quality of life at 3 months post-intervention | 13.48 (5.40) | 14.80 (6.33)
  Patient psychological quality of life at 2 weeks post-intervention | 28.58 (8.31) | 29.98 (5.99)
  Patient psychological quality of life at 3 months post-intervention | 28.66 (8.36) | 26.09 (8.27)
  Patient existential quality of life at 2 weeks post-intervention | 28.18 (5.35) | 28.15 (5.06)
  Patient existential quality of life at 3 months post-intervention | 28.25 (4.57) | 27.15 (4.83)
  Patient social quality of life at 2 weeks post-intervention | 24.59 (5.18) | 24.80 (5.32)
  Patient social quality of life at 3 months post-intervention | 25.28 (4.30) | 25.64 (3.51)
Statistical Analysis 1: Comparison: Acceptance and Commitment Therapy vs Education/Support; Test type: Superiority; p = 0.74, Mixed Models Analysis — P-value for study group x time interaction for patient physical quality of life. Two-tailed p-values <.05 were considered statistically significant; degrees of freedom = 76. Multiply imputed data were used; partial correlation = 0.06, 95% CI 2-sided [-0.25 to 0.38]
Statistical Analysis 2: Comparison: Acceptance and Commitment Therapy vs Education/Support; Test type: Superiority; p = 0.24, Mixed Models Analysis — P-value for study group x time interaction for patient psychological quality of life. Two-tailed p-values <.05 were considered statistically significant; degrees of freedom = 76. Multiply imputed data were used; partial correlation = 0.14, 95% CI 2-sided [-0.18 to 0.45]
Statistical Analysis 3: Comparison: Acceptance and Commitment Therapy vs Education/Support; Test type: Superiority; p = 0.78, Mixed Models Analysis — P-value for study group x time interaction for patient existential quality of life. Two-tailed p-values <.05 were considered statistically significant; degrees of freedom = 76. Multiply imputed data were used; partial correlation = 0.06, 95% CI 2-sided [-0.26 to 0.37]
Statistical Analysis 4: Comparison: Acceptance and Commitment Therapy vs Education/Support; Test type: Superiority; p = 0.29, Mixed Models Analysis — P-value for study group x time interaction for patient social quality of life. Two-tailed p-values <.05 were considered statistically significant; degrees of freedom = 76. Multiply imputed data were used; partial correlation = 0.13, 95% CI 2-sided [-0.19 to 0.44]

7. Secondary Outcome: PROMIS Global Health
Description: This 10-item measure assesses global health, including physical, mental, and social well-being. With the exception of pain, which is rated on a 0 to 10 scale, all items are rated on 5-point scales from 1 to 5. The item on pain is recoded from a 0-10 to a 1-5 scale and reverse-scored. Two additional items are reverse-scored. Then four of the items are summed, with higher physical quality of life subscale scores indicating better physical quality of life. Four other items are also summed with higher psychological quality of life subscale scores indicating better psychological quality of life. The subscale scores are converted to T-scores with a range from 16.2 to 67.7 for physical quality of life and a range from 21.2 to 67.6 for psychological quality of life. Higher T-scores for the physical and psychological quality of life subscales indicate a better outcome. The population mean for T-scores is 50 with a standard deviation of 10. This is a secondary outcome measure for caregivers.
Time Frame: 2 weeks and 3 months post-intervention
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Acceptance and Commitment Therapy | Education/Support
Number analyzed (Participants) | 20 | 20
T-score
  Caregiver physical quality of life at 2 weeks post-intervention | 46.11 (6.02) | 45.34 (5.24)
  Caregiver physical quality of life at 3 months post-intervention | 45.58 (4.42) | 44.68 (3.33)
  Caregiver psychological quality of life at 2 weeks post-intervention | 45.01 (5.11) | 43.48 (7.48)
  Caregiver psychological quality of life at 3 months post-intervention | 43.99 (4.50) | 43.30 (5.90)
Statistical Analysis 1: Comparison: Acceptance and Commitment Therapy vs Education/Support; Test type: Superiority; p = 0.92, Mixed Models Analysis — P-value for study group x time interaction for caregiver physical quality of life. Two-tailed p-values <.05 were considered statistically significant; degrees of freedom = 76. Multiply imputed data were used; partial correlation = 0.03, 95% CI 2-sided [-0.28 to 0.35]
Statistical Analysis 2: Comparison: Acceptance and Commitment Therapy vs Education/Support; Test type: Superiority; p = 0.79, Mixed Models Analysis — P-value for study group x time interaction for caregiver psychological quality of life. Two-tailed p-values <.05 were considered statistically significant; degrees of freedom = 76. Multiply imputed data were used; partial correlation = 0.06, 95% CI 2-sided [-0.26 to 0.37]

8. Secondary Outcome: Value Progress Subscale of the Valuing Questionnaire.
Description: This 5-item subscale assesses progress in living according to one's personal values, a construct related to activity engagement. Items are rated on 0 to 6 scales. The 5 items are summed with higher total subscale scores indicating greater progress in living according to one's personal values. The total subscale score range is 0 to 30. This is a secondary outcome measure for patients and caregivers.
Time Frame: 2 weeks and 3 months post-intervention
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acceptance and Commitment Therapy | Education/Support
Number analyzed (Participants) | 40 | 40
units on a scale
  Patient values progress at 2 weeks post-intervention: number analyzed (Participants) | 20 | 20
  Patient values progress at 2 weeks post-intervention | 21.71 (3.49) | 21.30 (5.29)
  Patient values progress at 3 months post-intervention: number analyzed (Participants) | 20 | 20
  Patient values progress at 3 months post-intervention | 22.71 (3.26) | 21.66 (5.09)
  Caregiver values progress at 2 weeks post-intervention: number analyzed (Participants) | 20 | 20
  Caregiver values progress at 2 weeks post-intervention | 23.05 (5.39) | 21.14 (4.33)
  Caregiver values progress at 3 months post-intervention: number analyzed (Participants) | 20 | 20
  Caregiver values progress at 3 months post-intervention | 22.97 (2.62) | 22.44 (3.05)
Statistical Analysis 1: Comparison: Acceptance and Commitment Therapy vs Education/Support; Test type: Superiority; p = 0.94, Mixed Models Analysis — P-value for study group x time interaction. Two-tailed p-values <.05 were considered statistically significant; degrees of freedom = 144. Multiply imputed data were used; partial correlation = 0.02, 95% CI 2-sided [-0.30 to 0.34]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected on each participant from the point of baseline until 21 weeks post-baseline.
Groups:
- Before Randomization: All-cause mortality and adverse events prior to randomization to a study arm
Arm/Group | Acceptance and Commitment Therapy | Education/Support | Before Randomization
All-Cause Mortality (participants affected / at risk) | 1/20 | 2/20 | 1/22
Serious Adverse Events (participants affected / at risk) | 1/20 | 2/20 | 1/22
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acceptance and Commitment Therapy (N=20) | Education/Support (N=20) | Before Randomization (N=22)
Deaths (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 1 (1) — All patients had advanced cancer at the time of enrollment and the serious adverse events (deaths) were expected and unrelated to the study intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/27/NCT04010227/Prot_SAP_000.pdf
  • Informed Consent Form: Consent Form for Patients (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/27/NCT04010227/ICF_001.pdf
  • Informed Consent Form: Consent Form for Family Caregivers (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/27/NCT04010227/ICF_002.pdf